CLINICAL TRIAL: NCT01843244
Title: Plethysmography as a Useful Intraoperative Monitor
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Justin M. Aden MD, University of Virginia Department of Anesthesiology
Other Study IDs: 15097
Record Dates: First submitted 2011-08-09; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Cardiovascular Diseases
Keywords: plethysmography
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Data from both the traditional invasive cardiac monitors and the Nonin will be collected simultaneously. The investigators will analyze Nonin data for peak and trough variation with respiration, area under the curve, time from trough to peak, and slope, and compare these to data collected from the invasive monitors to look for correlations in clinically important parameters such as blood pressure, central venous pressure, cardiac output, etc.

DETAILED DESCRIPTION:
After obtaining written consent to participate, the standard of care arterial line and PA catheter will be placed pre-operatively. The investigators will attach the Nonin pulse oximeter, as a second pulse oximeter probe, to patients undergoing surgical procedures which already require invasive cardiac monitors (arterial line, pulmonary artery catheter, etc). Data from both the traditional invasive cardiac monitors and the Nonin pulse oximeter will be collected as electronic files. Once both files are compiled they will be de-identified.

The investigators will also record medications and IV fluids given during surgery.

The Nonin Pulse Oximeter is clinically marketed for this indication

The investigators will analyze Nonin data for peak and trough variation with respiration, area under the curve, time from trough to peak, and slope, and compare these to data collected from the invasive monitors to look for correlations in clinically important parameters such as blood pressure, central venous pressure, cardiac output, etc.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older Patient scheduled for surgery that will have both an arterial catheter and a pulmonary artery catheter as standard of care Informed consent

Exclusion Criteria:

* Only the above inclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for surgery that will have both an arterial catheter and a pulmonary artery catheter as standard of care
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
waveform variation of the Nonin pulse oximeter compared with that of the arterial catheter | during surgery
  The investigators will analyze Nonin data for peak and trough variation with respiration, area under the curve, time from trough to peak, and slope, and compare these to data collected from the invasive monitors to look for correlations in clinically important parameters such as blood pressure, central venous pressure, cardiac output, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Thiele, MD, Principal Investigator — UVA Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States